CLINICAL TRIAL: NCT01987440
Title: Effect of Lubricating Gel for Pain Relief During Speculum Examination in Gynecologic Oncology Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erzincan Military Hospital (Other)
Responsible Party: Principal Investigator, Kemal GUNGORDUK, M.D, Erzincan Military Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: gungorduk16
Record Dates: First submitted 2013-11-12; First posted 2013-11-19 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain

ARMS (2):
- Lubricating Gel (Experimental): The speculum was warmed, and patients were informed about what was going to happen. The labia were spread from below to introduce the speculum, which was inserted at a 45-degree angle pointing downward then rotated horizontally as the insertion continued. A VAS score (insertion) was obtained at this point. Next, the bill of the speculum was opened up until the vaginal cuff could be seen, and the speculum was secured by turning the thumbnut. A second VAS score (dilation) was recorded. During speculum examination, cervical smear with cervical brush was obtained for pathologic assessment if necessary. The speculum was withdrawn slightly, which allowed the bill to close together, and at this stage (extraction) the final VAS score was obtained. In the gel group , a doctor placed 6,5 mL mL sterile lubricating gel on the top and bottom blades of the speculum. Length of the vagina was measured by the index finger.
  Interventions: Drug: lubricating gel
- water (Placebo Comparator): A VAS score (insertion) was obtained at this point. Next, the bill of the speculum was opened up until the vaginal cuff could be seen, and the speculum was secured by turning the thumbnut. A second VAS score (dilation) was recorded. During speculum examination, cervical smear with cervical brush was obtained for pathologic assessment if necessary. The speculum was withdrawn slightly, which allowed the bill to close together, and at this stage (extraction) the final VAS score was obtained. In the water group the speculum's top and bottom blades were moistened with 6,5 mL tap water previously loaded into a syringe kept at room temperature.After the speculum examination, pelvic examination was performed and length of the vagina (defined as distance from vaginal cuff to vaginal apex) was measured by the index finger.
  Interventions: Drug: lubricating gel

INTERVENTIONS:
Drug: lubricating gel

SUMMARY:
Pelvic examination, an important part of gynecologic oncology patients to help detect cancers recurrence or infections.Despite its importance, many women are reluctant and anxious about the procedure because of fear, as well as discomfort and pain. The objective of this study is to estimate whether using lubricating gel decreases patient pain during speculum insertion compared with using water in gynecologic oncology patients

ELIGIBILITY:
Inclusion Criteria:

*Female patients WHO came for surveillance for malignant gynecologic disease such as uterine cancer, cervix cancer, and ovarian cancer with or without radiotherapy and chemotherapy

Exclusion Criteria

* Women were undergoing Vulvectomy or Vaginectomy
* Women with narrow vagina for standard medium size of speculum for examination
* Women who underwent fertility sparing surgery.
* Women had vaginitis

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | During Speculum Examination Dilatation stage
  During Speculum Examination Dilatation stage

SECONDARY OUTCOMES:
visual analog scale insertion stage | uring Speculum Examination insertion stage
  During Speculum Examination insertion stage

OTHER OUTCOMES:
VAS score extraction | Durig extraction the speculum

CONTACTS AND LOCATIONS:
Locations (1):
- Tepecik Education and REserch Hospital, Izmir, Tepecik, Turkey (Türkiye)